CLINICAL TRIAL: NCT02053350
Title: Alanyl-glutamine Supplementation of Standard Treatment for C. Difficile Infection: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Alanyl-glutamine Supplementation of Standard Treatment for C. Difficile Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Cirle Warren, MD, Associate Professor, Department of Medicine, Infectious Disease, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17576; 17576 Protocol_Alanyl_Glutami (Other: UVA PI)
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; glutamine; diarrhea; alanyl-glutamine
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — alanylglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alanyl-glutamine (Experimental): Alanyl-glutamine, 44g, taken by mouth daily for 10 days.
  Interventions: Drug: Alanyl-glutamine

INTERVENTIONS:
Drug: Alanyl-glutamine — Alanyl-glutamine, 44g, taken by mouth daily for 10 days
  Other Names: alagln

SUMMARY:
The aim of this study is to test the efficacy of alanyl-glutamine supplementation in the treatment of C. difficile infection. We hypothesize that alanyl-glutamine when given with standard antibiotic treatment for C. difficile infection will decrease diarrhea, mortality and recurrent disease.

DETAILED DESCRIPTION:
This is a Phase II randomized, placebo-controlled, double-blinded, dose-ranging study to determine optimal effective dose and safety of AQ between 0, 4, 24, and 44 g doses administered orally for ten days concurrent with standard treatment (oral vancomycin at UVa) among first time incident cases of uncomplicated CDI in hospitalized persons age 50 and older. Our hypothesis is that AQ will reduce recurrence (primary outcome) and mortality (secondary outcome) at 60 days post-treatment. Furthermore, we hypothesize that alanyl-glutamine supplementation will be associated with decreased intestinal and systemic inflammation and improvement of intestinal microbial and metabolic profiles. We plan to enroll 260 patients, equally divided into 4 arms. Upon enrollment, participants will be randomized to either receive AQ at 4, 24, or 44 g or placebo (water). Study agent is administered once a day, orally or enterally, if feeding tube is present. Because we are enrolling subjects over a longer period of time, we will utilize block randomization to ensure that relative temporal balance is maintained throughout the trial. Participants will be followed up daily during treatment for adverse event monitoring and weekly for 60 days post-treatment for recurrences and survival. Blood, urine and stool specimens will be collected at days 0, 10 and 70 to assay for markers of inflammation and microbial and metabolic profiling.

The data set utilized for all initial baseline feature and demographic reporting will be the Intention to Treat Analysis Dataset, which will be comprised of all randomized participants. The primary dataset will be a Modified Intention to Treat Analysis Dataset for all endpoints, comprised of all participants who took at least one dose of study intervention (placebo or treatment), regardless of completeness of follow-up outcome data. The Safety Analysis Dataset will be all participants who took at least one dose of study intervention. The Per Protocol Analysis Dataset will be those patients who took at least 9 doses of study intervention for 9 days of the treatment period (10 days). Analysis will utilize ANOVA unless statistically significant differences in the distribution of baseline characteristics or features of non-normality are detected and relevant, at which point contingency utilization of ANCOVA, logistic regression, or other approaches as appropriate will be implemented. Treatment group level rates will be presented as incidence risk ratios relative to the control (placebo) group with 95% confidence intervals.

Safety endpoints will be evaluated on an individual AE by AE event via the DSMB and utilizing summary statistics during treatment and through duration of follow up. Adverse events will be presented by System Organ Class and will include information on start and stop date, severity, projected relationship, expectedness, and outcome and duration (the latter two after the event is considered to have concluded).

ELIGIBILITY:
Inclusion Criteria:

* Adult of either gender, 18 years or older, with C. difficile infection (CDI)
* Diarrhea associated with C. difficile positive stool assay
* Within 48 hours of receiving either metronidazole for mild-moderate disease or vancomycin for severe uncomplicated disease
* Admitted in the hospital at the time of enrollment
* Ability to provide informed consent
* Have an understanding of study procedures
* Ability to comply with study procedures for the entire length of the study

Exclusion Criteria:

* Hypotension or shock
* Megacolon or moderate to severe ileus
* Acute abdomen
* Severe leukocytosis (WBC > 20,000 cells /µL)
* Admission to intensive care unit on enrollment
* Inability to tolerate oral medication
* Other known etiology of diarrhea (e.g. other enteric pathogen, other intestinal disease)
* Inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
* Enrollment in another investigational drug trial
* Currently receiving other alternative treatment for CDI (e.g. antibiotics other than metronidazole or vancomycin; probiotics; immunoglobulin therapy; fecal transplant)
* Pregnancy
* Unavailable for follow-up visits
* Life expectancy of < 6 months
* Chronic liver disease or in subjects without known liver disease, ALT > 3x normal
* Chronic kidney disease or in subjects without known kidney disease, estimated Creatinine clearance of < 30 ml/min, even after rehydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cirle A. Warren, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alanyl-glutamine
Started | 7
Completed | 2
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Alanyl-glutamine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.86 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent C. Difficile Infection
Description: Day 40 clinical failure - clinical failure includes death or CDI recurrence assessed 40 days post randomization or lack of clinical cure
Time Frame: At day forty
Population: Number of Participants with Recurrent C. Difficile Infection
Measure: Count of Participants; unit: Participants
Arm/Group | Alanyl-glutamine
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Mortality
Description: Death from any cause at days 40, 70 and 190
Time Frame: Up to 6 months after end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Alanyl-glutamine
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months post randomization.
Description: All AEs including local and systemic reactions not meeting the criteria for "serious adverse events" will be captured on the appropriate CRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product
Arm/Group | Alanyl-glutamine
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alanyl-glutamine (N=7)
gastrointestinal symptoms (Gastrointestinal disorders) | 4 (4) — Vomiting Abdominal pain Diarrhea Nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02053350/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02053350/ICF_001.pdf